CLINICAL TRIAL: NCT00810524
Title: Influence of Antiviral Treatment to the Long-Term Prognosis of Patients With Chronic HBV Infection.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: The Third Affliated Hospital of Sun Yat-sen University, The Third Affliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU 5010 Hepatitis B
Record Dates: First submitted 2008-12-01; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; antiviral treatment; long term prognosis
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; Telbivudine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): 120 subjects (have family history of hepatic carcinoma or liver cirrhosis). Antiviral treatment are started when ALT is lower than 80u/L (early antiviral treatment).
  Interventions: Drug: lamivudine; Drug: Telbivudine; Drug: Enticavir; Drug: Adefovir Dipivoxil Tablets
- B (Active Comparator): 120 subjects (have family history of hepatic carcinoma or liver cirrhosis). Antiviral treatment are started when ALT is higher than 80u/L (regular antiviral treatment).
  Interventions: Drug: lamivudine; Drug: Telbivudine; Drug: Enticavir; Drug: Adefovir Dipivoxil Tablets
- C (Experimental): 180 subjects (have no family history of hepatic carcinoma or liver cirrhosis). Antiviral treatment are started when ALT is lower than 80u/L (early antiviral treatment).
  Interventions: Drug: lamivudine; Drug: Telbivudine; Drug: Enticavir; Drug: Adefovir Dipivoxil Tablets
- D (Active Comparator): 180 subjects (have no family history of hepatic carcinoma or liver cirrhosis). Antiviral treatment are started when ALT is higher than 80u/L (regular antiviral treatment).
  Interventions: Drug: lamivudine; Drug: Telbivudine; Drug: Enticavir; Drug: Adefovir Dipivoxil Tablets

INTERVENTIONS:
Drug: lamivudine — 100mg, P.O.,QD, duration: until HBeAg seroconversion for more than 2years.
Drug: Telbivudine — 600mg, P.O.,QD, duration: until HBeAg seroconversion for more than 2years.
Drug: Enticavir — 0.5mg, P.O.,QD, duration: until HBeAg seroconversion for more than 2 years.
Drug: Adefovir Dipivoxil Tablets — 10mg, P.O.,QD, duration: until HBeAg seroconversion for more than 2years.

SUMMARY:
Influence of antiviral treatment to the long term prognosis of patients with chronic HBV infection. The aim of antiviral treatment for HBV is to reduce the long term severe complications. In this study, the investigators divided patients with chronic HBV infection into two groups, which start early antiviral treatment and conventional antiviral treatment respectively. All the patients will be followed for ten years. From this study, the investigators want to find out the optimal time for patients with chronic HBV infection to start antiviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months.
* HBeAg positive.
* HBV DNA over 10E5 copies/ml.

Exclusion Criteria:

* Previous antiviral treatment for HBV.
* Co infection of HIV, HCV, HEV, HAV, or HAV.
* Evidence of hepatic carcinoma.
* Evidence of autoimmune disease.
* Evidence of thyroid disease.
* History of mental sickness.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
incidence rate of hepatic carcinoma | 10 years after treatment
incidence rate of liver cirrhosis | 10 years after treatment
incidence rate of fulminant hepatitis | 10 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gao zhiliang, M. D., Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (2):
- China (2):
  - The Third Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou, Guangdong